CLINICAL TRIAL: NCT00274027
Title: Randomised, Double-Blind, Placebo-Controlled, Cross-Over Study to Examine the Effects of Tiotropium on Lung Hyperinflation, Respiratory Mechanics and Dyspnea During Exercise in Patients With COPD
Brief Title: Mechanisms of Dyspnea Relief During Exercise in COPD Patients Following Treatment With Tiotropium (Spiriva)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.231
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium bromide

SUMMARY:
To explore the mechanisms of dyspnea relief during exercise in patients with COPD following treatment with tiotropium bromide (Spiriva)

DETAILED DESCRIPTION:
This was a single-centre, randomised, double-blind, placebo-controlled, cross-over study. The duration of subject participation was 9 weeks. There was an initial screening period of up to 2 weeks. The first screening visit consisted of medical history, clinical assessment, chronic dyspnea evaluation, complete pulmonary function testing, and a symptom-limited maximal incremental cycle exercise test. A second visit during the screening period was intended as a training of the subject to the procedures to be performed in the study, with specific focus on familiarisation with the constant work rate exercise test. The screening period was followed by 2 x 7 day treatment periods (1 x tiotropium and 1 x placebo), separated by a 4 week washout period. On the last day of each treatment period, the subject visited the clinic to complete a series of trial related procedures, including lung function measurements and a constant work rate exercise test at 75% Wcap to symptom limitation. Testing consisted of pulmonary function testing, dyspnea evaluation, and symptom-limited constant-load cycle exercise tests with measurements of cardiopulmonary parameters, symptom intensity and pulmonary mechanics. \

Study Hypothesis:

Dynamic hyperinflation restricts volume expansion during exercise and is suspected as a primary mechanism of dyspnea. The dissociation between drive or muscular effort to breathe and the mechanical response to increased volume (as reflected by an increased Pes/PImax: VT/predicted VC ratio) correlates well with the intensity of inspiratory difficulty during exercise in COPD. It was hypothesised that reduced Borg ratings at a standardized exercise level after tiotropium would correlate strongly with reduced restricted volume expansion during exercise (i.e., increased VT/IC and EILV/TLC ratios, and decreased IC and IRV). In other words, dyspnea and its predominant qualitative dimensions (i.e., inspiratory difficulty) result from patients being forced by DH to breathe at a high lung volume, at or above predicted TLC.

Comparison(s):

tiotropium bromide (Spiriva) vs. placebo

ELIGIBILITY:
Inclusion criteria: Patients with chronic obstructive pulmonary disease (COPD) with FEV1 < 70% predicted and FRC > 120% predicted, a cigarette smoking history > 20 pack-years, and moderate to severe chronic dyspnea

Exclusion criteria: patients with a history of asthma, allergic rhinitis or atopy; patients who participated in a rehabilitation program for COPD within 6 weeks prior to screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Borg dyspnea rating at a standardized exercise time (DyspneaSTD) during a constant work rate exercise challenge to symptom limitation at 75% maximal work capacity | up to 7 weeks

SECONDARY OUTCOMES:
Endurance time | up to 7 weeks
Borg leg discomfort | up to 7 weeks
Qualitative aspects of dyspnea | up to 7 weeks
Locus of sensory limitation | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Canada Ltd.
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Travers J, Laveneziana P, Webb KA, Kesten S, O'Donnell DE. Effect of tiotropium bromide on the cardiovascular response to exercise in COPD. Respir Med. 2007 Sep;101(9):2017-24. doi: 10.1016/j.rmed.2007.03.008. Epub 2007 May 1. PMID 17475459